CLINICAL TRIAL: NCT00035711
Title: VA HDL Intervention Trial (VA-HIT) Ancillary Study Data Analysis
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1008; R03HL069111 (NIH)
Record Dates: First submitted 2002-05-04; First posted 2002-05-06 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2005-11

CONDITIONS: Coronary Disease; Heart Diseases; Cardiovascular Diseases; Carotid Artery Diseases; Diabetes Mellitus, Non-insulin Dependent; Hypertension; Insulin Resistance; Obesity; Diabetes Mellitus
MeSH Terms: conditions — Coronary Disease; Heart Diseases; Cardiovascular Diseases; Carotid Artery Diseases; Diabetes Mellitus, Type 2; Hypertension; Insulin Resistance; Obesity; Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
To evaluate additional cardiovascular risk factors using data from the VA HDL Intervention Trial (VA-HIT).

DETAILED DESCRIPTION:
BACKGROUND:

The VA HDL Intervention trial (VA-HIT) was a multicenter, placebo controlled, randomized trial that showed that gemfibrozil significantly reduced major cardiovascular events in 2531 men with coronary heart disease, low levels of low density lipoprotein (LDL) cholesterol and low levels of high density lipoprotein (HDL) cholesterol. In addition to its unique lipid profile, the VA-HIT population also had a high prevalence of diabetes, impaired fasting glucose, or high fasting plasma insulin; central obesity; and hypertension, which are all components (together with high triglycerides and low HDL-cholesterol) of a constellation of risk factors known as the metabolic syndrome. Since prior clinical trials have not enrolled this type of population, the VA- HIT database is a unique resource.

DESIGN NARRATIVE:

The study used the VA-HIT database to study additional risk markers that were measured in the study population of 2,531 men with coronary heart disease. Specific analyses were: 1) the association between levels of glucose tolerance, insulin resistance and other features of the metabolic syndrome, occurrence of major cardiovascular outcomes, and gemfibrozil efficacy; 2) the effect of gemfibrozil on progression of carotid atherosclerosis, as measured by B-mode ultrasound; 3) the association between LDL particle size distribution and lipoprotein subclass distribution; homocysteine; lipoprotein(a); C-reactive protein, tissue plasminogen activator; fibrinogen; and factor VII; major cardiovascular outcomes and gemfibrozil efficacy.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-09; Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Rubins — VA Medical Center